CLINICAL TRIAL: NCT02136563
Title: oBservational Clinical Research In Chronic Kidney Disease Patients With Renal Anemia : Renal proGnosis in Patients With Hyporesponsive Anemia To Erythropoiesis Stimulating Agents, darbepoetiN Alfa
Brief Title: Renal Prognosis in Chronic Kidney Disease Patients With Hyporesponsive Anemia to Erythropoiesis Stimulating Agents
Acronym: BRIGHTEN
Status: Completed | Type: Observational
Sponsor: Translational Research Center for Medical Innovation, Kobe, Hyogo, Japan (Other)
Collaborators: Niigata University (Unknown)
Responsible Party: Sponsor
Other Study IDs: TRIGU1318; UMIN000013464 (Registry Identifier: UMIN-CTR)
Record Dates: First submitted 2014-05-07; First posted 2014-05-13 (Estimated); Last update posted 2020-06-18 (Actual); Status verified 2020-06

CONDITIONS: Renal Anemia; Chronic Kidney Disease
Keywords: Chronic kidney disease; Erythropoiesis stimulating agent response index; Hyporesponsive anemia to erythropoiesis stimulating agent; Observational study
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Darbepoetin alfa

SUMMARY:
This is an observational clinical research on patients with chronic kidney disease who are not on hemodialysis and receiving darbepoetin alfa to treat diagnosed renal anemia; the major objective is to explore novel erythropoiesis stimulating agent (ESA) response index in association with deterioration of renal function as well as occurrence of cardiovascular disease events.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are planning to start treatment with darbepoetin alfa within 8 weeks after enrollment,
2. Patients with eGFR <60 mL/min/1.73m2 at the latest examination performed within 8 weeks before enrollment,
3. Patients with a hemoglobin level <11.0 g/dL at the latest examination performed within 8 weeks before enrollment,
4. Patients aged at least 20 years or older at the time of providing informed consent,
5. Patients who voluntarily provided written informed consent to participate in the study.

Exclusion Criteria:

1. Patients who are planning to start hemodialysis or to have a renal transplant within 24 weeks after enrollment,
2. Patients with a history of treatment with ESA except the ones who were treated temporarily more than 12 weeks before the enrollment,
3. Patients with malignant tumor, hematological disease, or hemorrhagic lesions,
4. Patients with hypersensitivity to ESA or any ingredient thereof,
5. Pregnant, lactating or possibly pregnant women or those who wish to become pregnant during the study period,
6. Patients who are participating in other clinical study,
7. Patients who are assessed as not eligible for the study by the investigator.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic renal disease patients without dialysis who are diagnosed with renal anemia and are administered darbepoetin alfa at enrollment
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2014-04; Primary Completion 2019-08 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
Deterioration of renal function | For ninety six weeks after starting to administer darbepoetin alfa
Cardiovascular disease events | For ninety six weeks after starting to administer darbepoetin alfa

SECONDARY OUTCOMES:
Declination rate of estimated glomerular filtration rate(eGFR) | For ninety six weeks after starting to administer darbepoetin alfa
Safety assessment for every adverse event resulting from darbepoetin alfa administration | For ninety six weeks after starting to administer darbepoetin alfa

OTHER OUTCOMES:
Erythropoiesis resistance index (ERI) | For ninety six weeks after starting to administer darbepoetin alfa

CONTACTS AND LOCATIONS:
Overall Officials: Ichiei Narita, Principal Investigator — Niigata University Graduate School of Medicine
Locations (1):
- Niigata University Graduate School of Medicine, Niigata, Japan

REFERENCES:
- [Derived] Nakai K, Nishino T, Kagimura T, Narita I. Impact of transferrin saturation on cardiovascular events in non-dialysis-dependent chronic kidney disease patients treated with darbepoetin alfa. J Nephrol. 2024 Nov;37(8):2327-2335. doi: 10.1007/s40620-024-02000-y. Epub 2024 Jun 28. PMID 38941000